CLINICAL TRIAL: NCT06896552
Title: Investigating the Effect of Ketogenic Diet on Immunological Parameters in Advanced Cancer Patients Undergoing Immunotherapy
Brief Title: Single-Center Trial on Ketogenic Diet and Immunotherapy in Advanced Cancer This Study Evaluates the Safety and Effects of a Ketogenic Diet (KD) Combined With Immunotherapy in Adults With Advanced Melanoma, cSCC, or RCC.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Gal Markel, MD Ph.D. MBA, Deputy Director of Rabin Medical Center, and Director of Davidoff Center Rabin Medical Center, Full Professor of Clinical Microbiology & Immunology at the Sackler Faculty of Medicine, Tel Aviv University., Rabin Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0046-25-RMC
Record Dates: First submitted 2025-03-05; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Immunotherapy; Ketogenic Diet
Keywords: Metastatic Melanoma; Renal Cell Carcinoma; Ketogenic Diet; Dietary Intervention and Immunotherapy; Ketogenic diet (KD) and cancer treatment
MeSH Terms: conditions — Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Single-center, open-label, prospective, non-randomized, controlled, sequential two-arm clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic Diet (KD) Group: A high-fat, low-carb diet (intermittent schedule: 2 weeks on,1 week off)) (Experimental): Seven days (±2 days) before first dose of immunotherapy, patients will receive instructions to follow KD. The KD composition: 5-10% of the calories from carbohydrate, 20-30% protein and 60-70% fat. No calorie restriction will be applied, and patients will be instructed to eat to satiety. Supplemental MCT (medium chain triglyceride) oil or /and ketocal powder (Nutricia) will be added at the dietician's discretion in order to promote ketone production. During the period off the KD, the participants will be instructed to gradually follow standard diet composition (50-60% of the calories from carbohydrate, 15-20% protein and 20-30% fat). Diet protocol will be given to the patient along with specific menu suggestions for each individual.
  Interventions: Dietary Supplement: Ketogenic diet
- Standard Diet (SD) Group: A typical diet with no major changes. (No Intervention)

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — Ketogenic Diet as an Adjunct to Immunotherapy: Unlike many trials focused on chemotherapy or targeted therapies, this study specifically investigates the synergistic effects of the ketogenic diet with immune checkpoint inhibitors (ICIs), a promising approach for enhancing immunotherapy efficacy. The diet's high-fat, low-carbohydrate regimen is designed to shift metabolism towards ketone bodies and fatty acid utilization, potentially modulating immune responses and tumor immunogenicity in a way that standard diets do not.
  Arms: Ketogenic Diet (KD) Group: A high-fat, low-carb diet (intermittent schedule: 2 weeks on,1 week off))

SUMMARY:
This clinical trial aims to evaluate whether a ketogenic diet (KD), when combined with immunotherapy, can improve immune function and treatment outcomes in patients with advanced melanoma, cutaneous squamous cell carcinoma (cSCC), or renal cell carcinoma (RCC).

Why Is This Study Important? Immunotherapy is a promising cancer treatment, but not all patients respond well. Research suggests that diet, particularly a high-fat, low-carbohydrate ketogenic diet, may help boost the immune system and make treatments more effective.

What Will This Study Examine?

Researchers want to understand:

Is the ketogenic diet well-tolerated for cancer patients? Does the diet improve immune responses and treatment effectiveness?

How Will the Study Work?

Participants will be placed into one of two groups:

Ketogenic Diet (KD) Group: A structured high-fat, low-carb diet (intermittent schedule: 2 weeks on, 1 week off).

Standard Diet (SD) Group: A typical diet with no major changes. Throughout the study, a dietitian will closely support and guide you. Both groups will continue their standard immunotherapy treatment.

What Will Participants Do? Write their food intake three times a week to help assess dietary adherence Follow their assigned diet for 10 weeks Have weekly check-ins with a dietitian (in-person at the hospital or via phone) Have weekly blood glucose and ketone level checks using a home device. Provide monthly blood samples to measure immune response during routine immunotherapy infusions Provide stool samples for gut microbiome analysis at the start and end of the study Measure Monthly Weight, body composition, and resting calorie burn Complete quality-of-life questionnaires

What Are the Potential Benefits? Improved response to immunotherapy Better understanding of how diet influences cancer treatment Potential for a new supportive strategy for cancer care

This study may help uncover ways to enhance cancer treatment through personalized nutrition.

ELIGIBILITY:
Inclusion Criteria:

* • Males and females, age >= 18 years

  * Patients with a histologically confirmed melanoma or cSCC or RCC receiving first line treatment with combination nivolumab and ipilimumab /relatlimab or single agent ipilimumab, nivolumab, pembrolizumab, Cemiplimab.
  * Able to read, understand, and provide written informed consent
  * Willing and able to complete all study-specific procedures and visits
  * Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
  * Blood tests:

    * Creatinine (Cr) < 1.5 mg/dL.
    * Magnesium normal range ( 1.5 -2,6 mg/dL)
    * Liver function tests (LFTs) 2.5x upper limit of normal (ULN).
    * Neutrophils ≥ 1,000/mm3, platelets ≥ 50,000/mm3, Hb>8 g/dL
    * Women of childbearing potential must have a negative β-HCG pregnancy test documented within 1 week of registration.

Exclusion Criteria:

* • Individuals < 18 years of age

  * Unable or unwilling to provide consent
  * Other active malignancy (other than adequately treated and cured basal or squamous cell skin cancer, curatively treated in situ disease, or any other cancer from which the patient has been disease free >=2 years)
  * Currently consuming a low-carbohydrate (< 130 g/day) or KD or done so in the last 6-months
  * Patients currently participating in an interventional or therapeutic clinical trial involving the use of active anti-cancer therapy.
  * Active autoimmune diseases requiring active Immune suppressive medications
  * Systemic steroid therapy, excluding for replacement due to adrenal insufficiency
  * Major surgery within last 3 months
  * BMI <18 or >35
  * Medical contraindications to the intervention diet as determined by the treating physician.
  * Self-reported major dietary restrictions related to the intervention such as irritable bowel syndrome (IBS).
  * Patients with a history or active eating disorder
  * Uncontrolled Diabetes mellitus or patients receiving insulin
  * Known diagnosis of HIV
  * Known active hepatitis B or hepatitis C
  * Known inborn errors of lipid metabolism
  * Sever or uncontrolled Hyperlipidemia (total cholesterol over 400 mg / dL, low-density lipoprotein (LDL) above 300 mg / dL, triglycerides over 500 mg / dl.).
  * Pregnant or lactating.
  * Patients who have undergone a transplant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Adhering to the Ketogenic Diet and Experiencing Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to the end of treatment at 10 weeks
  This measure will assess the feasibility and tolerability of the ketogenic diet (KD) in cancer patients undergoing immunotherapy by evaluating:
  Diet Adherence: The number of participants who maintain KD for at least 80% of the study duration, based on dietary intake logs and ketone level measurements.
  Tolerability: The number of participants experiencing treatment-related adverse events (AEs), as assessed using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. The severity and frequency of AEs will be documented and categorized.
Change in Peripheral Blood Mononuclear Cell (PBMC) Composition at Baseline, During, and Post-Intervention | Monthly (week 0, 4, 10 ±1 week).
  This measure will evaluate changes in immune cell composition in response to the ketogenic diet (KD) and immunotherapy.
  PBMC Composition: Assessed using cytometry by time-of-flight (CyTOF) to characterize shifts in immune cell subsets (e.g., T cells, natural killer cells, monocytes).
  Data Analysis: Changes from the baseline will be reported as absolute values and fold-changes over time.
Serum Cytokine Levels at Baseline, During, and Post-Intervention | Monthly (week 0, 4, 10 ±1 week).
  This measure will evaluate changes in cytokine levels in response to the ketogenic diet (KD) and immunotherapy.
  Serum Cytokine Levels: Quantified using multiplex immunoassays to measure the concentrations of key cytokines, such as IL-2, IFN-γ, TNF-α, and IL-10.
  Data Analysis: Changes from baseline will be reported as absolute values and fold-changes over time.

SECONDARY OUTCOMES:
Overall response rate according to RECIST v1. | End of treatment at 10 weeks
Adherence to Dietary Interventions - Ketone Level Measurements | Weekly from Baseline (Week 0) to Week 10
  Ketone Level Measurements: Ketone levels will be measured to assess whether participants are in a state of ketosis (>0.3 Mm), indicating adherence to the ketogenic diet.
  Data Analysis: Ketone levels will be analyzed to determine adherence to the ketogenic diet.
Change in Body Weight (kg) Over the Study Period | Baseline (Week 0), Week 4, Week 10, and Week 14 (±1 week).
  Body weight (in kilograms) will be measured using a calibrated digital scale at specified time points. Changes from baseline will be reported as absolute weight differences and percentage change
Change in Quality of Life Score Assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | At enrollment (Baseline, Week 0) and at the end of treatment (Week 10).
  Quality of life will be assessed using the EORTC QLQ-C30 questionnaire, a validated tool for measuring cancer patients' health-related quality of life.
  The EORTC QLQ-C30 consists of 30 items, evaluating functional scales (physical, role, emotional, cognitive, and social functions), symptom scales (fatigue, pain, nausea/vomiting, etc.), and global health status.
  Scores range from 0 to 100. Higher scores on functional and global health scales indicate better quality of life.
  Higher scores on symptom scales indicate greater symptom burden (worse outcome).
  Changes from baseline to Week 10 will be reported as mean score differences.
Fecal microbiome | At enrollment (baseline) and at the end of treatment at 10 weeks
  Such as, but not limited to, 16S analysis
Sarcopenia | At enrollment (baseline) and at the end of treatment at 10 weeks
  Assessed using CT scans of the axial L3 sections and customized software
Body composition-- Fat Mass and Lean Mass | Monthly (week 0, 4, 10 ±1 week).
  This measure will assess changes in body composition using bioelectrical impedance analysis (BIA).
  Fat Mass(kg) and Lean Mass (kg): Body composition will be assessed using Bioelectrical Impedance Analysis (BIA) to measure fat mass(kg) and lean mass(kg).
  Data Analysis: Changes in fat mass and lean mass will be reported as absolute values and fold-changes over time.
Resting Energy Expenditure (REE) | Monthly (week 0, 4, 10 ±1 week).
  Measured by indirect calorimeter - Q-NRG
The Rate of immune-related adverse events | From enrollment to the end of treatment at 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] 1. Ribas A, Wolchok JD. Cancer immunotherapy using checkpoint blockade. Science. 2018;359(6382):1350-1355. 2. Hargadon KM, Johnson CE, Williams CJ. Immune checkpoint blockade therapy for cancer: An overview of FDA-approved immune checkpoint inhibitors. Int Immunopharmacol. 2018;62:29-39. 3. Haslam A, Prasad V. Estimation of the percentage of US patients with cancer who are eligible for and respond to checkpoint inhibitor immunotherapy drugs. JAMA Netw Open. 2019;2(5):e192535. 4. Golonko A, Pienkowski T, Swislocka R. Dietary factors and their influence on immunotherapy strategies in oncology: A comprehensive review. Cell Death Dis. 2024;15:254. 5. Weber DD, Aminzadeh-Gohari S, Tulipan J, Feichtinger RG. Ketogenic diet in cancer therapy. Aging (Albany NY). 2020;12(3):6018. 6. Klement RJ. The emerging role of ketogenic diets in cancer treatment. Curr Opin Clin Nutr Metab Care. 2017;20(1):28-34. 7. Harel M, Ortenberg R, Varanasi SK, Mangalhara KC, Mardamshina M, Markovits E, et al. Proteomics of melanoma response to immunotherapy reveals mitochondrial dependence. Cell. 2019;179:236-250.e218. 8. Ferrere G, Tidjani Alou M, Liu P, Goubet AG, Fidelle M, Kepp O, et al. Ketogenic diet and ketone bodies enhance the anticancer effects of PD-1 blockade. JCI Insight. 2021;6(2):e145207. 9. Jiang T, Zhou C, Ren S. Role of IL-2 in cancer immunotherapy. Oncoimmunology. 2016;5(6):e1163462. 10. Erickson N, Boscheri A, Linke B, Huebner J. Systematic review: Isocaloric ketogenic dietary regimes for cancer patients. Med Oncol. 2017;34(5):72. 11. Woolf EC, Curley KL, Liu Q, Scheck AC. The ketogenic diet alters the hypoxic response and affects expression of proteins associated with angiogenesis, invasive potential, and vascular permeability in a mouse glioma model. PLoS One. 2015;10:e0130357. 12. Weber DD, Aminzadeh-Gohari S, Tulipan J, Catalano L, Feichtinger RG, Kofler B. Ketogenic diet in the treatment of cancer - Where do we stand? Mol Metab. 2020;33:102-121. 13. Lussier DM, Woolf EC, Johnson JL, Brooks KS, Blattman JN, Scheck AC. Enhanced immunity in a mouse model of malignant glioma is mediated by a therapeutic ketogenic diet. BMC Cancer. 2016;16:310. 14. Rom-Jurek EM, Kirchhammer N, Ugocsai P, Ortmann O, Wege AK, Brockhoff G. Regulation of programmed death ligand 1 (PD-L1) expression in breast cancer cell lines in vitro and in immunodeficient and humanized tumor mice. Int J Mol Sci. 2018;19:563. 15. Husain Z, Huang Y, Seth P, Sukhatme VP. Tumor-derived lactate modifies antitumor immune response: Effect on myeloid-derived suppressor cells and NK cells. J Immunol. 2013;191:1486-1495. 16. Weber DD, Aminzadeh-Gohari S, Thapa M, Kofler B, Feichtinger RG. Ketogenic diets slow melanoma growth in vivo regardless of tumor genetics and metabolic plasticity. Cancer Metab. 2022;10:12. 17. Russo E, Nannini G, Amedei A. Exploring the food-gut axis in immunotherapy response of cancer patients. World J Gastroenterol. 2020;26(33):4919-4932. 18. Verhoog S, Taneri PE, Roa Diaz ZM, Marques-Vidal P, Troup JP, Bally L, et al. Dietary factors and modulation of bacteria strains of Akkermansia muciniphila and Faecalibacterium prausnitzii: A systematic review. Nutrients. 2019;11:1565. 19. Murphy S, Rahmy S, Gan D, Gao Y, Jiang H, Alves MR, et al. Ketogenic diet alters the epigenetic and immune landscape of prostate cancer to overcome resistance to immune checkpoint blockade therapy. Cancer Res. 2024;84(10):1597-1612. 20. Zhang Y, Kurupati R, Liu L, Zhou XY, Zhang G, Hudaihed A, et al. Enhancing CD8(+) T cell fatty acid catabolism within a metabolically challenging tumor microenvironment increases the efficacy of melanoma immunotherapy. Cancer Cell. 2017;32:377-391.e379. 21. NutRatio.com NutRatio [Internet]. [cited 2022 Nov 24]. Available from: https://nutratio.com/ 22. Römer M, Dörfler J, Huebner J. The use of ketogenic diets in cancer patients: A systematic review. Clin Exp Med. 2021;21(4):501-536